CLINICAL TRIAL: NCT00987935
Title: A Multicenter, Open Label, Phase I/Randomized II Study to Evaluate Safety, Pharmacokinetics and Efficacy of BIBF 1120 in Comparison With Sorafenib for Advanced Hepatocellular Carcinoma Patients in Asia.
Brief Title: A Phase I / II Trial of Nintedanib in Asian Hepatocellular Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.39
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; nintedanib

ARMS (2):
- Nintedanib (BIBF 1120) (Experimental): Phase I dose escalation and phase II using dose determined in phase I
  Interventions: Drug: BIBF 1120
- Sorafenib (Active Comparator): Twice daily dosing in phase II
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400 mg twice daily
  Arms: Sorafenib
Drug: BIBF 1120 — Twice daily
  Arms: Nintedanib (BIBF 1120)

SUMMARY:
This study is to evaluate the safety, appropriate dose, and efficacy of BIBF 1120 in liver cancer patients

ELIGIBILITY:
Inclusion criteria:

1. Hepatocellular carcinoma, either histologically/cytologically confirmed or clinically diagnosed, which is not amenable to curative surgery or loco-regional therapy
2. Age 18 years or older
3. Eastern Cooperative Group performance score of 2 or less
4. Child-Pugh score of 7 or less
5. Written informed consent in accordance with International Conference on Harmonisation (ICH) and Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

1. Prior systemic therapy for metastatic/unresectable hepatocellular carcinoma (for phase II)
2. More than one line of prior systemic therapy for metastatic/unresectable hepatocellular carcinoma (for phase I)
3. Uncontrolled or refractory ascites to adequate medical therapy
4. Bilirubin greater than 1.5 times upper limit of normal
5. Aspartate amino transferase or alanine amino transferase greater than 5 times upper limit of normal
6. Absolute neutrophil count less than 1500/microliter
7. Platelet count less than 75000/microliter
8. Hemoglobin less than 9 g/dL
9. Serum creatinine greater than 1.5 times upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-10; Primary Completion 2014-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- South Korea (6):
  - 1199.39.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.39.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.39.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.39.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.39.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1199.39.82006 Boehringer Ingelheim Investigational Site, Seoul
- Taiwan (10):
  - 1199.39.88606 Boehringer Ingelheim Investigational Site, Changhua
  - 1199.39.88609 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1199.39.88610 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1199.39.88605 Boehringer Ingelheim Investigational Site, Taichung
  - 1199.39.88602 Boehringer Ingelheim Investigational Site, Tainan
  - 1199.39.88608 Boehringer Ingelheim Investigational Site, Tainan
  - 1199.39.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1199.39.88603 Boehringer Ingelheim Investigational Site, Taipei
  - 1199.39.88604 Boehringer Ingelheim Investigational Site, Taoyuan
  - 1199.39.88607 Boehringer Ingelheim Investigational Site, Yunlin County

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial consisted of 2 Phases. Patients were stratified into 1 of 2 groups according to their aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and Child-Pugh score at baseline.
Pre-assignment Details: Group 1 patients had a baseline Child-Pugh score of 5 or 6, and AST (aspartate aminotransferase ) and ALT (alanine transaminase) ≤2 times the upper limit of normal (ULN).
  Group 2 patients had a baseline Child-Pugh score of 7, or AST or ALT >2 to ≤5 times ULN
Groups:
- Phase I Group I, 100 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the maximal tolerated dose (MTD) and pharmacokinetics (PK) of nintedanib.
- Phase I Group 1, 150 mg Nintedanib Bid; Phase I Group 2, 150 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD and pharmacokinetics (PK) of nintedanib.
- Phase I Group 1, 200 mg Nintedanib Bid; Phase I Group 2, 200 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD and pharmacokinetics (PK) of nintedanib.
- Phase I Group 2, 50 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 50 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD and pharmacokinetics (PK) of nintedanib.
- Phase I Group 2, 100 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the MTD and pharmacokinetics (PK) of nintedanib.
- Phase II, 200 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules twice daily (bid).
  Phase II: Patients were randomly assigned to open-label treatment with nintedanib or sorafenib. Patients were stratified for macro-vascular invasion (MVI) and/or extra-hepatic spread (EHS).
- Phase II, 400 mg Sorafenib Bid: Oral administration of Sorafenib 400 mg film coated tablets twice daily (bid).
  Phase II: Patients were randomly assigned to open-label treatment with nintedanib or sorafenib. Patients were stratified for macro-vascular invasion (MVI) and/or extra-hepatic spread (EHS).
Period: Overall Study
Arm/Group | Phase I Group I, 100 mg Nintedanib Bid | Phase I Group 1, 150 mg Nintedanib Bid | Phase I Group 1, 200 mg Nintedanib Bid | Phase I Group 2, 50 mg Nintedanib Bid | Phase I Group 2, 100 mg Nintedanib Bid | Phase I Group 2, 150 mg Nintedanib Bid | Phase I Group 2, 200 mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Started | 4 | 3 | 3 | 3 | 7 | 3 | 16 | 63 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 (On-treatment at analysis cut-off date (16 July 2014).) | 1 (On-treatment at analysis cut-off date (16 July 2014).) | 0
Not Completed | 4 | 3 | 3 | 3 | 7 | 3 | 15 | 62 | 32
Not completed — Progressive disease | 3 | 2 | 3 | 2 | 5 | 3 | 9 | 48 | 23
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 10 | 6
Not completed — Refused to continue taking trial med. | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 4 | 2
Not completed — Reason other than those specified above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): Treated set included all patients who received at least one dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Group I, 100 mg Nintedanib Bid | Phase I Group 1, 150 mg Nintedanib Bid | Phase I Group 1, 200 mg Nintedanib Bid | Phase I Group 2, 50 mg Nintedanib Bid | Phase I Group 2, 100 mg Nintedanib Bid | Phase I Group 2, 150 mg Nintedanib Bid | Phase I Group 2, 200 mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 3 | 16 | 63 | 32 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.5) | 55.7 (4.2) | 47.7 (6.8) | 64.3 (15.3) | 62.3 (11.1) | 68.7 (10.1) | 56.1 (11.7) | 58.2 (12.6) | 61.2 (11.5) | 58.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 6 | 16
  Male | 4 | 3 | 3 | 3 | 7 | 2 | 13 | 57 | 26 | 118

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose in Phase I
Description: The MTD was defined as the highest dose studied for which the incidence of DLTs was 0/3 or less than 2/6 patients during the first treatment course.
Time Frame: 4 weeks
Population: Treated set (Patients from the dose escalation part that were not replaced for MTD determination)
Measure: Number; unit: mg
Groups:
- Group 1; Group 2: Patients treated with nintedanib belonging to Group1 from the 2 phases,
  Phase I Group 1 treatment consists of nintedanib, 100, 150 or 200 mg twice daily (bid)
  Phase II treatment consists of Nintedanib 200 mg twice daily (bid)
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 9 | 15
mg | 200 | 200

2. Primary Outcome: Time to Progression (TTP) in Phase II
Description: TTP according to Response Evaluation Criteria in Solid Tumours (RECIST) 1.0 criteria based on central independent review. TTP RECIST 1.0 was defined as the time from randomisation to disease progression according to RECIST 1.0.
Time Frame: From randomization until data cut-off (28 Sep 2012); Up to 77 weeks
Population: Treated set, only phase II participants.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 63 | 32
months | 2.73 [0.99 to 5.55] | 3.71 [1.77 to 7.36]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 1.357, 95% CI 2-sided [0.802 to 2.296] — Hazard ratio from Cox proportional hazards model stratified by macroscopic vacular invasion, extrahepatic spread, or both present vs both absent. HR below 1 favors Nintedanib

3. Secondary Outcome: Time to Progression (TTP) in Phase II (Follow-up Analyses)
Description: as for outcome 2
Time Frame: From randomization until disease progression or data cut-off (16 Jul 2014); Up to 171 weeks
Population: Treated set, Only phase II participants
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 63 | 32
months | 2.76 [0.99 to 5.55] | 3.71 [1.77 to 7.36]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 1.213, 95% CI 2-sided [0.730 to 2.014] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Incidence and Intensity of Adverse Events (AEs) Reported as the Number of Patients With AEs According to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 Throughout the Treatment Period.
Description: Incidence and worst intensity (severity) of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: AEs with an onset during therapy with study treatment or within 28 days after discontinuation of study treatment (up to 1066 days)
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Phase I Group I, 100 mg Nintedanib Bid | Phase I Group 1, 150 mg Nintedanib Bid | Phase I Group 1, 200 mg Nintedanib Bid | Phase I Group 2, 50 mg Nintedanib Bid | Phase I Group 2, 100 mg Nintedanib Bid | Phase I Group 2, 150 mg Nintedanib Bid | Phase I Group 2, 200 mg Nintedanib Bid | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 7 | 3 | 16 | 63 | 32
participants
  Grade 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 12 | 1
  Grade 2 | 2 | 2 | 1 | 0 | 0 | 1 | 4 | 15 | 4
  Grade 3 | 2 | 1 | 1 | 1 | 3 | 2 | 5 | 17 | 18
  Grade 4 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 8 | 5
  Grade 5 | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 10 | 4

5. Secondary Outcome: Incidence of Dose Limiting Toxicity in Phase I
Description: Number of patients with dose limiting toxicity are presented
Time Frame: 4 weeks
Population: Treated set (Phase I patients from the dose escalation part that were not replaced for MTD determination).
Measure: Number; unit: participants
Groups:
- Phase I Group 1, 100 mg Nintedanib Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid).
  Phase I: A standard 3+3 dose escalation part to determine the maximal tolerated dose (MTD) and pharmacokinetics (PK) of nintedanib.
Arm/Group | Phase I Group 1, 100 mg Nintedanib Bid | Phase I Group 1, 150 mg Nintedanib Bid | Phase I Group 1, 200 mg Nintedanib Bid | Phase I Group 2, 50 mg Nintedanib Bid | Phase I Group 2, 100 mg Nintedanib Bid | Phase I Group 2, 150 mg Nintedanib Bid | Phase I Group 2, 200 mg Nintedanib Bid
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3 | 3
participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Objective Tumour Response by RECIST
Description: Objective RECIST 1.0 tumour response was defined as Complete Response (CR) or Partial Response (PR) and was derived from the patient's best objective RECIST 1.0 response based on central independent review.
  95% Confidence Interval presented below are computed by Clopper and Pearson method.
Time Frame: From randomization until data cut-off (16 July 2014); Up to 171 weeks
Population: Treated set, only phase II participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 63 | 32
percentage of participants | 6.3 [1.8 to 15.5] | 3.1 [0.1 to 16.2]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS by RECIST 1.0 was defined as the duration from date of randomisation to date of progression or death, whichever occurred earlier, based on central independent review.
Time Frame: From randomization until data cut-off (16 July 2014); Up to 171 weeks
Population: Treated set, only phase II participants.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 63 | 32
months | 2.66 [0.99 to 5.55] | 3.71 [1.77 to 7.36]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 1.186, 95% CI 2-sided [0.728 to 1.932] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration from date of randomisation to the date of death.
Time Frame: From randomization until data cut-off (16 July 2014); Up to 171 weeks
Population: Treated set, include only phase II participants
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Phase II, 200 mg Nintedanib Bid | Phase II, 400 mg Sorafenib Bid
Number analyzed (Participants) | 63 | 32
months | 10.18 [5.19 to 16.85] | 10.71 [7.29 to 16.66]
Statistical Analysis 1: Comparison: Phase II, 200 mg Nintedanib Bid vs Phase II, 400 mg Sorafenib Bid; Test type: Superiority or Other; Hazard Ratio (HR) = 0.940, 95% CI 2-sided [0.593 to 1.489] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: AUC0-12,ss,Norm (Area Under the Plasma Concentration-time Curve Between 0 and 12 Hours at Steady State, Normalised Values) of Nintedanib
Description: AUC0-12,ss,norm (area under the plasma concentration-time curve between 0 and 12 hours at steady state, normalised values) of Nintedanib
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: Pharmacokinetic set (PKS): The PK set was a subset of the treated set and included all patients who received at least one dose of trial medication and for whom at least one PK observation was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Groups:
- Group 2: Phase I Group 2 treatment consists of nintedanib, 50, 100, 150 or 200 mg twice daily:
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
(ng*h/mL)/mg | 1.97 (97.1) | 3.82 (64.1)

10. Secondary Outcome: AUC0-12,ss,Norm (Area Under the Plasma Concentration-time Curve Between 0 and 12 Hours at Steady State, Normalised Values) of BIBF 1202 (Metabolite of Nintedanib)
Description: AUC0-12,ss,norm (area under the plasma concentration-time curve between 0 and 12 hours at steady state, normalised values) of BIBF 1202 (metabolite of Nintedanib).
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
(ng*h/mL)/mg | 3.50 (157) | 8.95 (114)

11. Secondary Outcome: AUC0-12,ss,Norm (Area Under the Plasma Concentration-time Curve Between 0 and 12 Hours at Steady State, Normalised Values) of BIBF 1202 Glucuronide (Metabolite of Nintedanib)
Description: AUC0-12,ss,norm of BIBF 1202 glucuronide (Metabolite of Nintedanib):
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
(ng*h/mL)/mg | 16.9 (144) | 45.0 (124)

12. Secondary Outcome: Cmax,ss,Norm (Maximum Concentration of the Nintedanib in Plasma at Steady State, Normalised Values)
Description: Cmax,ss,norm (maximum concentration of the Nintedanib in plasma at steady state, normalised values).
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 22 | 23
(ng/mL)/mg | 0.348 (98.8) | 0.630 (68.9)

13. Secondary Outcome: Cmax,ss,Norm (Maximum Concentration of the BIBF 1202 in Plasma at Steady State, Normalised Values)
Description: Cmax,ss,norm (maximum concentration of the BIBF 1202 in plasma at steady state, normalised values).
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 22 | 23
(ng/mL)/mg | 0.519 (148) | 1.01 (118)

14. Secondary Outcome: Cmax,ss,Norm (Maximum Concentration of the BIBF 1202 Glucuronide in Plasma at Steady State, Normalised Values)
Description: Cmax,ss,norm (maximum concentration of the BIBF 1202 glucuronide in plasma at steady state, normalised values).
  Detailed time points of sampling are:
  Phase I and selected phase II patients in the Nintedanib arm:
  Cycle 1, Day 15 to 16: Immediately prior to swallowing the dose of nintedanib (predose) and 1 hour (h), 2 h, 3 h, 4 h, 5 h, 7 h, 10 h, 12 h and 24 h after drug administration on Day 15; Cycle 2, Day 1: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 1; Cycle 2, Day 15: Immediately prior to swallowing the dose of nintedanib (predose) and 2 h after drug administration on Day 15.
Time Frame: Day1, Day15 and Day 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)/mg
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 22 | 23
(ng/mL)/mg | 1.56 (139) | 3.48 (139)

15. Secondary Outcome: fe0-12,ss (Fraction Excreted in Urine Between 0 and 12 Hours at Steady State) for Nintedanib
Description: fe0-12,ss (fraction excreted in urine between 0 and 12 hours at steady state) for Nintedanib.
  The reported value corresponds to the percentage of administered dose.
Time Frame: 0 to 4 hours (h), 4 to 12 h, and 12 to 24 h after nintedanib
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 22 | 23
percentage | 0.227 (94.6) | 0.286 (46.0)

ADVERSE EVENTS:
Time Frame: AEs with an onset during therapy with study treatment or within 28 days after discontinuation of study treatment (up to 1066 days)
Groups:
- Phase I Group I Nintedanib, 100 mg Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid) for the Group I patients during Phase I
- Phase I Group I Nintedanib, 150 mg Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid) for the Group I patients during Phase I
- Phase I Group I Nintedanib, 200 mg Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules twice daily (bid) for the Group I patients during Phase I
- Phase I Group II Nintedanib, 50 mg Bid: Oral administration of Nintedanib (BIBF 1120) 50 mg soft gelatine capsules twice daily (bid) for the Group II patients during Phase I
- Phase I Group II Nintedanib, 100 mg Bid: Oral administration of Nintedanib (BIBF 1120) 100 mg soft gelatine capsules twice daily (bid) for the Group II patients during Phase I
- Phase I Group II Nintedanib, 150 mg Bid: Oral administration of Nintedanib (BIBF 1120) 150 mg soft gelatine capsules twice daily (bid) for the Group II patients during Phase I
- Phase I Group II Nintedanib, 200 mg Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules twice daily (bid) for the Group II patients during Phase I
- Phase II Nintedanib, 200 mg Bid: Oral administration of Nintedanib (BIBF 1120) 200 mg soft gelatine capsules twice daily (bid) during Phase II
- Phase II Sorafenib, 400 mg Bid: Oral administration of Sorafenib 400 mg film coated tablets twice daily (bid) during Phase II
Arm/Group | Phase I Group I Nintedanib, 100 mg Bid | Phase I Group I Nintedanib, 150 mg Bid | Phase I Group I Nintedanib, 200 mg Bid | Phase I Group II Nintedanib, 50 mg Bid | Phase I Group II Nintedanib, 100 mg Bid | Phase I Group II Nintedanib, 150 mg Bid | Phase I Group II Nintedanib, 200 mg Bid | Phase II Nintedanib, 200 mg Bid | Phase II Sorafenib, 400 mg Bid
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 0/3 | 3/3 | 4/7 | 1/3 | 10/16 | 29/63 | 18/32
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 7/7 | 3/3 | 16/16 | 61/63 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Group I Nintedanib, 100 mg Bid (N=4) | Phase I Group I Nintedanib, 150 mg Bid (N=3) | Phase I Group I Nintedanib, 200 mg Bid (N=3) | Phase I Group II Nintedanib, 50 mg Bid (N=3) | Phase I Group II Nintedanib, 100 mg Bid (N=7) | Phase I Group II Nintedanib, 150 mg Bid (N=3) | Phase I Group II Nintedanib, 200 mg Bid (N=16) | Phase II Nintedanib, 200 mg Bid (N=63) | Phase II Sorafenib, 400 mg Bid (N=32)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visceral arterial ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Group I Nintedanib, 100 mg Bid (N=4) | Phase I Group I Nintedanib, 150 mg Bid (N=3) | Phase I Group I Nintedanib, 200 mg Bid (N=3) | Phase I Group II Nintedanib, 50 mg Bid (N=3) | Phase I Group II Nintedanib, 100 mg Bid (N=7) | Phase I Group II Nintedanib, 150 mg Bid (N=3) | Phase I Group II Nintedanib, 200 mg Bid (N=16) | Phase II Nintedanib, 200 mg Bid (N=63) | Phase II Sorafenib, 400 mg Bid (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 3 | 12 | 5
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 11 | 7
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Eye discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3 | 0 | 3 | 18 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 1 | 1 | 2 | 11 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 14 | 11
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 13 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 5 | 3 | 6 | 28 | 18
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 2 | 7 | 19 | 4
Plicated tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 5 | 19 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 3
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 5 | 14 | 4
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 3
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 11 | 4
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 12 | 6
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 2 | 0 | 1 | 1 | 2 | 7 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 2 | 0 | 2 | 0 | 4 | 9 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 6 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Haematocrit increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 2 | 1 | 8 | 25 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 4 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 8 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 2 | 1 | 0 | 3 | 9 | 6
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 3 | 3
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 9 | 4
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 18 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 10 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 5 | 10 | 9
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights